CLINICAL TRIAL: NCT00308451
Title: "A Randomized, Double Blinded, Placebo Controlled, Parallel Arm, Study to Evaluate the Improvement in Glycemic Control After Daily Administration of Chromium Picolinate and Biotin in Patients With Type 2 Diabetes Mellitus"
Brief Title: A 30 Day Acute Efficacy and Safety Study of Chromium Picolinate + Biotin on Glycemic Control in Overweight or Obese Subjects With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition 21, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N21 CPB-03001
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2006-03-29 (Estimated); Status verified 2006-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: chromium; chromium picolinate; type 2 diabetes mellitus; fructosamine; glycemic control; OGTT
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — picolinic acid; Biotin

INTERVENTIONS:
Drug: Chromium Picolinate (600 mcg Cr+3) + biotin (2 mg)

SUMMARY:
The purpose of the proposed work is to assess the effects of a dietary supplement, containing chromium (600 mcg per day) provided by chromium picolinate and biotin (2 mg per day) on glycemic control in type 2 diabetes. Specifically, this study will assess whether use of the supplement will lower the post-prandial rise in blood glucose experienced after ingestion of a 75g carbohydrate load, relative to placebo, in type 2 diabetic patients. The study will also assess the chronic effects of supplementation over a 4-week period (relative to placebo) on fasting plasma levels of glucose, insulin, lipids and lipoproteins.

DETAILED DESCRIPTION:
The purpose of this work is to assess the effects of a dietary supplement, containing chromium (600 mcg per day) provided by chromium picolinate and biotin (2 mg per day) on glycemic control in type 2 diabetes who are currently taking an oral antidiabetic agent (OAD) and failing therapy with OADs. Subjects entering the trial must have a HbA1c >/= 7.0% and have an OGTT >/= 200 mg/dL at 2 hours post consumption of a 75 g glucose beverage. The study is an acute 30 day intervention in conjunction with the subject's current OADs and standard of care in comparison to placebo.

Specifically, this study will assess whether use of the supplement will lower the post-prandial rise in blood glucose experienced after ingestion of a 75g carbohydrate load, relative to placebo, in type 2 diabetic patients as measured by the area under the curve for glucose (AUCg). The study will also assess the acute effects of supplementation over a 4-week period (relative to placebo) on fasting plasma levels of glucose, fructosamine, insulin, lipids and lipoproteins.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes > 12 months.
2. Post-prandial blood glucose (glucose > 200 mg/dl) levels consistent with an ADA diagnosis of diabetes as confirmed during the screening visit.
3. Male and female between the ages of 18 and 65 years.
4. HbA1c > 7.0%.
5. Use of treatment regimens including diet and exercise and/or drug therapy for diabetes are allowed. Drug therapy may include alpha-glucosidase inhibitors (e.g. acarbose, voglibose, miglitol) and oral hypoglycemic agents such as sulfonylureas and metformin and thiazolidinediones (TZDs). Insulin use is not allowable
6. No changes in medication dosage within 60 days prior to entering trial.
7. Subjects with a body mass index (BMI) >25 and < 35.
8. Fasting triglycerides < 400. [32]
9. Willing to complete all study related requirements.
10. Subject will provide written consent to participate in the trial and this consent must be given voluntarily.

Exclusion Criteria:

1. Diagnosis of type I diabetes.
2. Hypoglycemic event requiring EMS intervention < 12 months.
3. Diabetic Ketoacidosis (DKA) < 12 months.
4. Subjects taking any supplement containing chromium within the previous 90 days prior toenrollment.
5. Creatinine > 2.0 x ULN; AST or ALT > 2.0 x ULN; Total Bilirubin > 1.5 x ULN.
6. COPD, CHF, Angina, HTN, MI, or any other CVD requiring hospitalization within the previous 12 months.
7. History of cerebrovascular accident (CVA), pulmonary embolism (PE), or an unresolved deep vein thrombosis (DVT).
8. History of CABG, PTCA, or any other reperfusion therapy < 12 months.
9. Uncontrolled high blood pressure (seated: systolic > 160 mmHg or diastolic > 90 mmHg)
10. History of any serious immunosuppressive disorder or undergoing current immunosuppressive therapy.
11. Female subjects who are pregnant or nursing, or are planning on becoming pregnant during the study. No hormone replacement therapy for post-menopausal subjects.
12. Hepatic disease, impaired thyroid, or impaired renal function, or other diseases known to affect glucose or lipid metabolism. TSH must be within range of normality to enter trial.
13. Diagnosed or self-reported alcoholism or substance-abuse problems
14. Any psychiatric or mental health issue that would prevent the subject from completing the study
15. Any illness or complication factor that, in the opinion of the investigator, would jeopardize the subject's health or well being by participating in the study or would interfere with the subject successfully completing the study.
16. Current participation in any other clinical research trial for any product or device, or participation in said clinical trials within 30 days prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-11; Study Completion 2004-04

PRIMARY OUTCOMES:
Primary(baseline versus final): AUCg as recorded from a 2-hour OGTT with 75 g glucose beverage; fructosamine; fasting plasma glucose.

SECONDARY OUTCOMES:
Secondary (baseline versus final): Lipid panels (Total-C, HDL, LDL, VLDL), lipid ratios , apolipoprotein A and B.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Geohas, MD, Principal Investigator — Radiant Research - Chicago
Locations (1):
- Radiant Research Chicago, Chicago, Illinois, United States